CLINICAL TRIAL: NCT06654401
Title: Electrical Cardioversion As a Predictor in Postoperative Preservation of Sinus Rhythm in Patients with Persistent Atrial Fibrillation Before Radio Frequency Pulmonary Vein Isolation
Brief Title: Electrical Cardioversion As a Predictor in Postoperative Preservation of Sinus Rhythm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Shmatov Dmitry, Deputy Director (Cardiac Surgery), Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECPV-CSP-0723
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Persistent
Keywords: Atrial Fibrillation; Cardioversion; Catheter ablation; Late recurrence; Left atrial voltage; Left atrial volume
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-center study with 2 groups of patients (investigating and control arms)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency pulmonary vein isolation in patients with previous electrical cardioversion (Experimental): Depending on the duration of atrial fibrillation and anatomic parameters of the left atrium (according to heart ultrasound), patients will undergo electric cardioversion before the primary radiofrequency catether pulmonary veins' isolation. The experimental group will be subdivided into a persistent AF patients who were successfully cardioverted in sinus rhythm and persistent AF patients who failed to restore sinus rhythm during DC at the time of catheter ablation.
  Interventions: Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: 24-hour ECG Monitor; Procedure: Electroanatomic mapping
- Radiofrequency pulmonary vein isolation in patients without previous electrical cardioversion (Active Comparator): Primary interventional treatment is performed without restoration of the sinus rhythm.
  Interventions: Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: 24-hour ECG Monitor; Procedure: Electroanatomic mapping

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Standard assessment of the parameters of the left atrium: size, volume, volume indices
Diagnostic Test: 24-hour ECG Monitor — Assessment of cardiac arrhythmias according to 24-hour monitoring data
Procedure: Electroanatomic mapping — Intraoperative assessment of low voltage areas (potential fibrosis zones)

SUMMARY:
The aim of this study is to evaluate benefits of electric cardioversion in the early and long-term postoperative period in patients after radiofrequency catheter isolation of pulmonary veins. Parameters of the left atrium will be evaluated by transthoracic echocardiography and electroanatomic mapping. Preservation of the sinus rhythm will be assessed by 24-hour electrocardiographic monitoring.

The main question that is planned to be answered is:

Does a reverse remodeling of the left atrium and/or a decrease in the progression of the fibrosis zone occur after performing electrical cardioversion (and before subsequent catheter ablation) in patients with persistent and long-standing persistent atrial fibrillation (AF)? Can performed electrical cardioversion serve as a predictor of AF freedom in this group of patients?

Participants will undergo a follow-up examinations (echocardiography, ECG, 24-hour ECG monitoring) at the 3rd, 6th and 12th months after catheter ablation. Based on the results of these examinations, the recurrence rate of AF will be estimated.

Two groups of patients will include both persistent and long-standing persistent AF. Experimental group will include patients who underwent electrical cardioversion before the intervention, and active comparator group will include those patients who did not undergo it. The experimental group will be subdivided into a persistent AF patients who were successfully cardioverted in sinus rhythm and persistent AF patients who failed to restore sinus rhythm during DC at the time of catheter ablation. Analysis and comparison of subgroups will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the patient to participate in the study.
* Persistent atrial fibrillation resistant to antiarrhythmic drugs for 6 months or more
* The size of the left atrium is less than 55 mm, volume is less than 130 ml, volume index (LP) is less than 55 ml/m2

Exclusion Criteria:

* Reversible causes of atrial fibrillation (hyperthyroidism, pericarditis, myocarditis).
* Patients in need of myocardial revascularization and/or heart valvular disease correction.
* Any previous intervention (including MAZE surgery, thoracoscopic ablation; implanted occluder of the auricle of the left atrium.).
* Patients with severe concomitant pathology requiring correction.
* Contraindications for administration of anticoagulant therapy.
* Documented presence of a blood clot in the cavity of the left atrium or other reasons preventing the insertion of catheters into the left atrium.
* BMI of 40 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation 6 months after catheter ablation | Echocardiographic assessment of the parameters of the left atrium and 24-hour ECG monitoring is performed at the time of admission to the hospital; after 3,6 and 12 months after intervention or the latest data in the event of death, whenever comes first
  Absence of events of sustained atrial tachycardia according to 24-hour ECG monitoring

SECONDARY OUTCOMES:
Reverse remodeling of the left atrium and improvement of the contractility of the left ventricle | Echocardiographic assessment of the parameters of the left atrium and 24-hour ECG monitoring is performed at the time of admission to the hospital; after 3,6 and 12 months after intervention or the latest data in the event of death, whenever comes first
  An increase in the LV ejection fraction, a decrease in the volume and size of the left atrium according to transthoracic echocardiography
Freedom from atrial fibrillation 12 months after catheter ablation | Echocardiographic assessment of the parameters of the left atrium and 24-hour ECG monitoring is performed at the time of admission to the hospital; after 3,6 and 12 months after intervention or the latest data in the event of death, whenever comes first
  Absence of events of sustained atrial tachycardia according to 24-hour monitoring
Improving the quality of life of patients with atrial fibrillation | Patients fill out questionnaires upon admission to the hospital; 3, 6 and 12 months after surgical treatment or the latest data in the event of death, whenever comes first
  Assessment of the quality of life of patients with atrial fibrillation based on a questionnaire:
  Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire - provides an overall score; plus scores for symptoms, daily activities, treatment concerns, and treatment satisfaction.
  Overall or subscale scores range from 0-100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Clinic, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not planned to be shared with other parties

REFERENCES:
- [Background] Kamada H, Mori K, Ueda N, Wakamiya A, Nakajima K, Kamakura T, Wada M, Ishibashi K, Yamagata K, Inoue Y, Miyamoto K, Nagase S, Noda T, Izumi C, Noguchi T, Kusano K, Aiba T. Impact of Pre-Ablation Direct Current Cardioversion for Persistent Atrial Fibrillation to Predict Recurrence of Atrial Fibrillation after Catheter Ablation. Int Heart J. 2022;63(5):828-836. doi: 10.1536/ihj.22-135. PMID 36184544
- [Background] Kang JH, Lee DI, Kim S, Kim MN, Park YM, Ban JE, Choi JI, Lim HE, Park SW, Kim YH. Prediction of long-term outcomes of catheter ablation of persistent atrial fibrillation by parameters of preablation DC cardioversion. J Cardiovasc Electrophysiol. 2012 Nov;23(11):1165-70. doi: 10.1111/j.1540-8167.2012.02339.x. Epub 2012 Aug 8. PMID 22882453
- [Background] Choi SH, Yu HT, Kim D, Park JW, Kim TH, Uhm JS, Joung B, Lee MH, Hwang C, Pak HN. Late recurrence of atrial fibrillation 5 years after catheter ablation: predictors and outcome. Europace. 2023 May 19;25(5):euad113. doi: 10.1093/europace/euad113. PMID 37099677
- [Background] Hanaki Y, Machino-Ohtsuka T, Aonuma K, Komatsu Y, Machino T, Yamasaki H, Igarashi M, Sekiguchi Y, Nogami A, Ieda M. Preprocedural restoration of sinus rhythm and left atrial strain predict outcomes of catheter ablation for long-standing persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2020 Jul;31(7):1709-1718. doi: 10.1111/jce.14540. Epub 2020 May 16. PMID 32391641
- [Background] Lizewska-Springer A, Dabrowska-Kugacka A, Lewicka E, Drelich L, Krolak T, Raczak G. Echocardiographic predictors of atrial fibrillation recurrence after catheter ablation: A literature review. Cardiol J. 2020;27(6):848-856. doi: 10.5603/CJ.a2018.0067. Epub 2018 Jun 20. PMID 29924375